CLINICAL TRIAL: NCT01609335
Title: Normative Values for Cognitive Testing and Alzheimer's Imaging Biomarkers in Young Adults (30-49yo)
Brief Title: Normative Values for Cognitive Testing and Alzheimer's Imaging Biomarkers in Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Val Lowe, Consultant - Diagnostic Radiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-006972
Record Dates: First submitted 2012-05-23; First posted 2012-05-31 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitively Normal Subjects (Other): Study participation will consist of tests of memory and thinking, a MRI, and two PET scans. F-18 FDG and C-11 Pittsburgh compound B (PiB) are two drugs used in PET scans.
  Interventions: Drug: F-18 FDG; Drug: C-11 PiB

INTERVENTIONS:
Drug: F-18 FDG — One time intravenous administration of 17 millicurie (mCi) +/- 10%
Drug: C-11 PiB — One time intravenous administration of 10-20 mCi

SUMMARY:
Biomarkers of Alzheimer's disease (AD) occupy an essential place in recently formulated diagnostic criteria for AD where their role is to identify the pathophysiological processes underlying cognitive impairment or to predict time to dementia. Three of these biomarkers are brain imaging tests (amyloid PET, fludeoxyglucose (FDG) PET, and structural MRI). In order to effectively use AD biomarkers for diagnostic and prognostic purposes, continuous values much be divided into normal and abnormal ranges. This requires that a cut point(s) be established in the continuous distribution of values for each biomarker.

The investigators objective in this proposal is to obtain imaging biomarker data in a group of individuals who are appropriate for establishing normative values for AD biomarkers. The investigators believe the most valid approach to establishing biomarker cut points is to base them on the upper bound of the range observed in young to early-middle-age subjects in whom the presence of occult AD pathology is extremely unlikely. Based on a large volume of community-based autopsy data, that upper age limit would be about 50 years old. The lower age bound for a group of subjects used to establish normative AD biomarker values would have to be based on considerations of brain maturation, which may continue into the middle- to late-20s. Thus, taking the above into consideration, the ideal age range for establishing normative AD imaging biomarker data (amyloid PET, FDG PET, and structural MRI) may be ages 30-49 years old.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal males or females aged 30 to 49 years old.

Exclusion Criteria:

1. Subjects unable to lie down without moving for up to 45 minutes.
2. Women who are pregnant or cannot stop breast feeding for 24 hours.
3. Claustrophobic patients unable to tolerate the scans (no sedation can be offered).
4. Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Normal values for amyloid PET, FDG and Magnetic Resonance Imaging | 2 days
  Biomarkers of Alzheimer's disease (AD) occupy an essential place in recently formulated diagnostic criteria for AD where their role is to identify the pathophysiological processes underlying cognitive impairment or to predict time to dementia. Three of these biomarkers are brain imaging tests (amyloid PET, FDG PET, and structural MRI). In order to effectively use AD biomarkers for diagnostic and prognostic purposes, continuous values much be divided into normal and abnormal ranges. This requires that a cut point(s) be established in the continuous distribution of values for each biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Josie Williams, BS, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States